CLINICAL TRIAL: NCT02410434
Title: Examining Performance Ethnography as a Lesbian, Gay , Bisexual and Transgender (LGBT) Stigma Reducing Strategy in Swaziland and Lesotho
Brief Title: Reducing Lesbian, Gay , Bisexual and Transgender (LGBT) Stigma in Swaziland and Lesotho
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Carmen Logie, MSW, PhD, Assistant Professor, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: #30344
Record Dates: First submitted 2015-03-30; First posted 2015-04-07 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Social Stigma
Keywords: Stigma; lesbian; gay; bisexual; transgender
MeSH Terms: conditions — Social Stigma; Homosexuality, Female; Homosexuality; Bisexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LGBT Stigma Reduction Intervention (Experimental): Participants will complete a pre-test, followed by a performance ethnography where they will watch theatre performances that illustrate stigma experienced by LGBT persons in Swaziland and Lesotho. They will have the opportunity to participate in these theatre performances to demonstrate reduced stigma and increased acceptance of LGBT persons. They will then complete a post-test, followed by a 6 week follow up survey.
  Interventions: Other: LGBT Stigma Reduction Intervention

INTERVENTIONS:
Other: LGBT Stigma Reduction Intervention — Participants will complete a pre-test, followed by a performance ethnography where they will watch theatre performances that illustrate stigma experienced by LGBT persons in Swaziland and Lesotho. They will have the opportunity to participate in these theatre performances to demonstrate reduced stigma and increased acceptance of LGBT persons. They will then complete a post-test, followed by a 6 week follow up survey.

SUMMARY:
The specific objectives of this study are reduce stigma towards lesbian, gay, bisexual, and transgender persons in Swaziland and Lesotho, using performance ethnography at community roundtables.

DETAILED DESCRIPTION:
This project aims to develop performance ethnography approaches to reduce stigma towards lesbian, gay, bisexual and transgender (LGBT) persons in Swaziland and Lesotho by holding performance ethnography at community roundtables in Swaziland and Lesotho.

This project involved a critical ethnography with in-depth individual interviews conducted with LGBT communities in Swaziland and Lesotho. Following this, the investigators conducted a performance ethnography that involved: a) presenting theatre specialists and PRAs with the qualitative data; b) working together to highlight narratives, themes and visual images from this data; c) developing scripts for participatory theatre performances; d) implementing the theatre performances at community roundtables, with participants completing a pre and post-test and 6 week follow up.

The investigators will implement 2 interconnected KTE strategies in each location (Swaziland, Lesotho): (1) participatory theatre (PT) training/development and (2) community roundtables. (1) Participatory theatre (PT) training with SGM: The investigators will engage 6 SGMY (2 MSM, 2 WSW, 2 transgender) as PRA in each location. PRA will work with a theatre specialist to develop 3 short plays to highlight lived experiences of a) stigma and discrimination and b) resilience among MSM, WSW and trans persons. PRA will undertake a 4-week PT training program, including: PT processes; assessing. Phase 1 data; developing scenes; and production. PRA will work with community animators who will perform the scenarios to protect the privacy of the PR.

The investigators will implement community roundtables are to: a) raise awareness of SGM issues and b) reduce stigma. Purposive sampling will be employed to engage diverse stakeholders. Roundtables, 2 hours in duration, will be cofacilitated by PRA. The aim is to conduct 2 meetings in Swaziland and 2 in Lesotho, each with 20-25 participants, including groups identified as key to SGM wellbeing in Phase 1 (e.g. educators; law enforcement; civil society; LGBTQ groups). Community animators will enact the 3 plays developed by SGM using PT techniques. Plays will address narratives of stigma and discrimination that emerge in Phase 1 among SGM participants. Community animators will perform each play once to illustrate the situation and problem; the story will culminate in a crisis with no solution offered. Each play will be performed a second time, and roundtable participants can 'stop' the action at any point where there is a challenge. The participant that 'stops' the play will come up and replace the character and depict a possible solution or 'intervention.

To evaluate the project's outcomes the investigators will conduct cross-sectional surveys with roundtable participants (n=100) who will complete a pre/post-test evaluation and 6 week follow up. The primary outcome will be measured using the 'Attitudes Towards Lesbians and Gay Men Scale' (ATLG-R) to assess changes in phobia, stigma and knowledge regarding SGM issues following the participatory theatre event. The survey will also include questions about attitudes towards HIV related stigma. Socio-demographic information will be collected from all survey participants including age, gender, highest level of education, nationality, marital status, current household income, type of work, number of children, and religion. MANOVA will be used to assess pre/post-test differences across variables.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 18 years of age or older for being able to give informed consent and be willing to complete a follow up survey.

Exclusion Criteria:

* Participants who are 17 years of age or younger were exuded for not being able to give informed consent.
* Participants who were unwilling to complete a follow up survey were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2015-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Attitudes towards lesbian and gay men scale | 3 months
  assesses attitudes and stereotypes regarding LGBT persons

SECONDARY OUTCOMES:
HIV-related stigma | 3 months
  attitudes towards people living with HIV
Civic participation | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Logie, PhD, Principal Investigator — University of Toronto, Factor-Inwentash Faculty of Social Work
Locations (2):
- Southern Africa Nazarene University, Manzini, Eswatini
- Maluti School of Nursing, Maseru, Lesotho